CLINICAL TRIAL: NCT00001088
Title: A Phase I Safety and Immunogenicity Trial of the Facilitated HIV-1 Gag-Pol DNA Vaccine (APL-400-047, Apollon, Inc.) Given Intramuscularly by Needle and Syringe or Biojector 2000 Needle-Free Jet Injection System in HIV-1 Uninfected Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Rona Siskind, DAIDS
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 031
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-09-29 (Estimated); Status verified 2008-09

CONDITIONS: HIV Infections
Keywords: Injections, Intramuscular; AIDS Vaccines; HIV Seronegativity; Dose-Response Relationship, Immunologic; Fusion Proteins, gag-pol; Vaccines, DNA; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections | interventions — Bupivacaine

INTERVENTIONS:
Biological: APL 400-047
Drug: Bupivacaine hydrochloride

SUMMARY:
To evaluate the safety, tolerability and immunogenicity in humans of the APL-400-047 vaccine when administered intramuscularly by needle and syringe at 1 of 3 doses or by Biojector at the intermediate dose. [AS PER AMENDMENT 07/98: To evaluate the tolerability, safety, and immunogenicity of an increased dose in an additional group of volunteers.] DNA-based immunization mimics live-attenuated virus vaccination by stimulation of both the humoral and cellular arms of the immune system; thus, potentially providing the advantages of a live virus vaccination but without the potential risks. It is essential that novel vaccine strategies (including DNA-based immunizations) continue to be developed and enter Phase I human testing because to date, no candidate vaccine from any of the approximately 30 AVEG Phase I or II trials has progressed to a Phase III efficacy trial. Use of a Biojector jet gun for vaccine delivery may also have potential psychological, comfort, safety and immunologic advantages over the traditional needle and syringe method of delivery.

DETAILED DESCRIPTION:
DNA-based immunization mimics live-attenuated virus vaccination by stimulation of both the humoral and cellular arms of the immune system; thus, potentially providing the advantages of a live virus vaccination but without the potential risks. It is essential that novel vaccine strategies (including DNA-based immunizations) continue to be developed and enter Phase I human testing because to date, no candidate vaccine from any of the approximately 30 AVEG Phase I or II trials has progressed to a Phase III efficacy trial. Use of a Biojector jet gun for vaccine delivery may also have potential psychological, comfort, safety and immunologic advantages over the traditional needle and syringe method of delivery.

A total of 40 volunteers receive four immunizations each (at months 0, 1, 2 and 6) as follows:

10 volunteers are enrolled at the 100 microgram dose given intramuscularly (IM) by needle and syringe. If this dose appears safe and well tolerated through Day 14, 20 more volunteers are enrolled at the 300 microgram dose; 10 receiving vaccine administered by needle and syringe, 10 receiving vaccine administered by Biojector. If the 300 microgram dose appears safe and well tolerated through Day 14 in the 10 volunteers who receive intramuscular (IM) injections with needle and syringe, an additional group of volunteers are enrolled at the 1000 microgram dose given with needle and syringe. NOTE: Within each group of 10 volunteers, 8 receive APL-400-047, 2 receive control preparation (bupivacaine carrier alone). [AS PER AMENDMENT 07/98: An additional group of 12 volunteers will be treated at a dose of 3000 micrograms administered by needle and syringe. Ten of these volunteers will receive APL-400-047 formulated with bupivacaine as a facilitating agent; the remaining 2 patients will receive control preparation (bupivacaine carrier alone).] [AS PER AMENDMENT 4/27/99: Volunteers previously primed with either 300 or 1000 micrograms of the APL-400-047 vaccine receive an additional dose of DNA (or control, for control volunteers in the original protocol) followed one month later by two monthly canarypox (or placebo for control volunteers in the original protocol) boosts.]

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Negative ELISA for HIV within 8 weeks of immunization.
* CD4 count >= 400 cells/mm3.
* Normal history and physical examination.
* Negative for Hepatitis B surface antigen.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions and symptoms are excluded:

* Positive for anti-dsDNA antibodies.
* Medical or psychiatric condition or occupational responsibilities that preclude compliance with the protocol.
* Present psychosis.
* Active syphilis (eligible if serology documented to be a false positive or due to remote, i.e., > 6 months treated, infection).
* Active tuberculosis (eligible if positive purified protein derivative test and normal chest x-ray showing no evidence of TB and not requiring isoniazid therapy).

Concurrent Medication:

Excluded:

* Immunosuppressive medications.

Patients with the following prior conditions are excluded:

* History of immunodeficiency, chronic illness, or autoimmune disease.
* History of cancer unless there has been surgical excision followed by a sufficient observation period to give a reasonable assurance of cure.
* History of suicide attempts, recent suicidal ideation or past psychosis.
* History of anaphylaxis or other serious adverse reactions to vaccines.
* History of severe allergic reaction to any substance, requiring hospitalization or emergent medical care (e.g., Stevens-Johnson syndrome, bronchospasm, or hypotension).
* Hypersensitivity to bupivacaine or other amide-type anesthetics.

Prior Medication:

Excluded:

* Prior receipt of HIV-1 vaccines or placebo recipient in a previous HIV vaccine trial.
* Use of experimental agents within 30 days prior to study.
* Live attenuated vaccines within 60 days of study.
* Medically indicated subunit or killed vaccines (e.g., influenza, pneumococcal) within 2 weeks prior to study.

Prior Treatment:

Excluded:

Receipt of blood products or immunoglobulin in the past 6 months.

Risk Behavior:

Excluded:

Volunteers having identifiable higher risk behavior for HIV infection as determined by screening questions designed to identify risk factors for HIV infection, specifically:

* History of injection drug use within the last 12 months prior to enrollment.
* Higher or intermediate risk sexual behavior as defined by the AVEG (i.e., meeting the criteria for AVEG Risk Group C or D).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40
Dates: Start 1997-07; Primary Completion 2001-02 (Actual); Study Completion 2001-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mulligan M, Study Chair
Locations (4):
- United States (4):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Univ of Rochester Med Ctr, Rochester, New York
  - Vanderbilt Univ Hosp, Nashville, Tennessee
  - Univ of Washington / Pacific Med Ctr, Seattle, Washington

REFERENCES:
- [Background] Goepfert P, Mulligan M, Corey L, Graham B, Evans T, Weinhold K, Stablein D, Ginsberg R. AVEG 031: phase I evaluation of a gag-pol facilitated DNA vaccine for HIV-1 prevention. Int Conf AIDS. 1998;12:635 (abstract no 33216)
- [Background] Tellez I, Sabbaj S, Bansal A, Goepfert P, Evans T, Graham B, Ginsberg R, Weiner D, Corey L, Weinhold K, Mulligan M. HIV-specific T-cell responses in seronegative volunteers immunized with an HIV-1 gag-pol DNA vaccine. 7th Conference on Retroviruses and Opportunistic Infections. 2000 Jan 30-Feb 2 (abstract no 656)